CLINICAL TRIAL: NCT06842875
Title: Effect of a Technology-based Collaborative Model on Persistent Hypertension and Preventive Care Attendance Among Postpartum People With Hypertensive Disorders of Pregnancy
Brief Title: Rhode Island - Statewide Postpartum Hypertension Remote Surveillance
Acronym: RI-SPHERES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: Brown University (Other); Kent Hospital, Rhode Island (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2184383
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-02

CONDITIONS: Hypertension in Pregnancy; Postpartum Preeclampsia; Postpartum Complication
Keywords: postpartum hypertensive disorders of pregnancy; postpartum preeclampsia; digital health; collaborative care model; population health; self-measured blood pressure
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Both remote hypertension monitoring programs are managed by a different nurse practitioner who, by necessity, will not be masked. However, all care providers who provide perinatal care for enrolled participants will be masked to their patient's study group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RI-SPHERES (Experimental): A technology enabled collaborative care model. Participants will receive a LTE-enabled blood pressure (BP) cuff that syncs to a smartphone application (app) to send automated reminders and provide adaptive messaging tailored to distinct BP values and symptoms. The first six weeks of the program will focus on BP control, and the remaining time will help transition people to receive recommended preventive care. As part of the collaborative care model, the nurse practitioner will lead weekly meetings with a multidisciplinary clinical team about all enrolled people.
  Interventions: Behavioral: RI-SPHERES
- Standard self-measured blood pressure program (Active Comparator): Our hospital has a remote hypertension monitoring program that recommends daily blood pressure ascertainment for 6 weeks, at which time they are discharged and provided printed resources to encourage preventive care in the next few months. In this program, patients manually enter their self-measured BPs into the electronic medical record for the clinical team to manually review and respond.
  Interventions: Behavioral: Standard self-measured blood pressure program

INTERVENTIONS:
Behavioral: RI-SPHERES — Participants assigned to the RI-SPHERES group will be introduced virtually or in-person to the care manager (CM), who demonstrate how to communicate directly with patients through the app for medical or non-medical needs. Each participant will learn how to obtain SMBP, sync the LTE-enabled BP cuff to the RI-SPHERES app, and respond to adaptive messaging pertaining to BP measurements, which include the ability to receive on-demand education on postpartum topics (e.g., HDP, breastfeeding, mood disorders) per participant preference. During the study period, the CM will respond to needs elicited from the SDoH screening by facilitating referrals to community resources. After six weeks, the focus of RI-SPHERES will transition to preventive care in addition to SMBP. The CM will engage monthly with each study participant to ensure they have a primary care provider and to facilitate preventive care visits or specialist appointments, if needed.
  Arms: RI-SPHERES
Behavioral: Standard self-measured blood pressure program — Participants assigned to the routine care group meet virtually or in-person with a member of WIH's existing SMBP program and enroll in WIH's EPIC MyChart Portal to allow the SMBP program to receive patient-entered BP measurements and respond to messages. Participants will be provided with BP cuffs and taught how to obtain SMBP and report their BP through MyChart. At six weeks postpartum, WIH SMBP staff send a MyChart message to recommend BP ascertainment once per month and to describe the importance of attending a clinical visit with a primary care provider within a year of birth.
  Arms: Standard self-measured blood pressure program

SUMMARY:
This is a hybrid type 1 non-inferiority implementation effectiveness trial among postpartum patients with hypertension (N=1536) that will test the hypothesis that RI-SPHERES (a technologically enabled collaborative care model) is non-inferior to a standard self-measured blood pressure program in terms of persistent hypertension at six weeks postpartum and preventive care receipt within one year of delivery.

DETAILED DESCRIPTION:
Uncontrolled hypertensive disorders of pregnancy (HDP) are a major source of maternal mortality. National guidelines recommend blood pressure (BP) measurement 3-10 days after discharge and ≥1 preventive care visit within one year of delivery. Yet, barriers such as childcare or transportation issues reduce adherence to in-person BP checks, particularly among racial or ethnic minority patients. Programs in which patients self-measure BP (SMBP) at home show promising results regardless of patient race. However, a recent meta-analysis concluded current SMBP programs do not reduce maternal mortality or racial disparities in clinical outcomes, potentially due to their specific limitations: they end within six weeks of birth (though HDP can persist for months) and have decreased engagement with non-White people or those living in disadvantaged areas, though these populations are at the highest risk of persistent HTN and its adverse long-term effects. Thus, there is an urgent need to optimize SMBP programs to target short- and long-term HDP-related morbidity and to broadly implement these programs to eliminate disparities in HDP-related outcomes. One such program is Rhode Island (RI)-Statewide Postpartum HypErtension REmote Surveillance (RI-SPHERES), a technology-based SMBP program that aims to reduce short- and long-term HDP-associated morbidity in RI using the collaborative care model, a health services intervention that improves health outcomes and reduces racial disparities on a population level for people with chronic conditions. The proposed research aims to determine the effectiveness of RI-SPHERES in reducing short- and long-term morbidity associated with HDP throughout RI. This builds upon our pilot RCT (NCT05595629), in which a standard SMBP program was compared to a SMBP program that used a Bluetooth-enabled BP cuff that syncs to a smartphone application (app) to send automated reminders and provide adaptive messaging tailored to distinct BP values and symptoms. RI-SPHERES will expand this SMBP program to provide app-based patient-informed educational content on HDP-specific preventive care and bidirectional communication with RI-SPHERES staff for one year postpartum. Incorporating adaptive and automatic messaging increases RI-SPHERES' scalability by reducing clinical staff burden. However, formal analysis of factors that may hinder widespread implementation of RI-SPHERES is needed. Thus, we will conduct a Hybrid Type I Non-Inferiority Implementation-Effectiveness Trial among 1536 patients with HDP that compares a standard SMBP program to RI-SPHERES in terms of persistent HTN at six weeks postpartum and receipt of preventive care within one year of delivery (Specific Aim 1). We will examine the effect of both programs on increasing equity in terms of race, ethnicity, language, and geography for postpartum patients with HDP in Rhode Island (Specific Aim 2). We will also develop an implementation toolkit to facilitate the dissemination of RI-SPHERES (Specific Aim 3). The proposed project is expected to deliver a mechanism that will fill multiple research gaps for HDP identified by the US Preventive Services Task Force: 1) addressing health inequities through multilevel interventions, 2) evaluating SMBP programs; and 3) mitigating HDP's short- and long-term health consequences of HDP.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum patient aged 18 years or more at any birthing hospital in Rhode Island
* Diagnosed during pregnancy or after delivery with hypertensive disorder of pregnant
* English-, Spanish-, Portuguese-, or Haitian-Creole-speaking
* Smartphone ownership

Exclusion Criteria:

* Prior enrollment in this trial
* Prisoners or incarcerated people
* Inability or unwillingness to provide informed consent
* Inability to communicate with study team, despite an interpreter

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1536 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Persistent hypertension | Six weeks postpartum
  Persistent stage II hypertension will be defined as systolic blood pressure of 140 mmHg or higher and/or diastolic blood pressure of 90 mmHg or higher

SECONDARY OUTCOMES:
Attendance of preventive care visit | From six weeks postpartum until one year postpartum
  Participant attends a non-urgent appointment during which an internal medicine physician, family medicine physician, or primary care advanced practice provider (APP, including nurse practitioners or physician assistants) ascertains BP and provides patient counseling pertaining to HTN. While obstetrician-gynecologists (OBGYNs) or certified nurse midwives (CNMs) can provide preventive care, for this aim, visits provided by an OBGYN or CNM will only qualify if the visit occurs ≥6 weeks postpartum and the medical record states that HTN was discussed in the visit.
Blood pressure ascertainment | 1-10 days after hospital discharge
  Participant measured any BP (either in-person or via self-measured blood pressure)
Total number of self-measured blood pressure assessments provided to program in immediate postpartum period | Hospital discharge to six weeks postpartum
  Number of blood pressures sent in to the participant's self-measured blood pressure program (RI-SPHERES or standard program)
Total number of self-measured blood pressure assessments provided to program after six weeks postpartum | Six weeks postpartum until one year postpartum
  Number of blood pressures sent in to the participant's self-measured blood pressure program (RI-SPHERES or standard program)
Severe maternal morbidity after hospital discharge | Hospital discharge until 6 weeks postpartum
  Severe maternal morbidity, as defined by the Centers for Disease Control's composite.
Persistent stage I hypertension | Six weeks, six months, and 12 months postpartum
  Systolic blood pressure between 130-139 mmHg and/or diastolic blood pressure between 80-89 mmHg
Persistent stage II hypertension | Six and 12 months postpartum
  Systolic blood pressure at or above 140 mmHg and/or diastolic blood pressure at or above 90 mmHg
Severe hypertension after hospital discharge | Hospital discharge to 6 weeks postpartum
  Systolic blood pressure at or above 160 mmHg or diastolic blood pressure at or above 110 mmHg on two or more occasions
Emergency room visit for hypertension-related etiology | Hospital discharge to 6 weeks postpartum
  Presentation to emergency room for hypertension-related chief complaint
Readmission to inpatient hospital for hypertension-related etiology | Hospital discharge until 6 weeks postpartum
  Readmission to inpatient hospital for hypertension-related chief complaint
Initiation or titration of antihypertension medication | Hospital discharge to 6 weeks postpartum
  Initiation or increase in dose titration of antihypertensive medication(s)
Postpartum visit attendance | Four to six weeks postpartum
  Attendance to the recommended in-person postpartum visit
System usability scale | Six weeks, six months, and 12 months postpartum
  A 10-question survey designed to provide a global view of subjective assessments of usability for a technology-based program or intervention
Client satisfaction questionnaire | Six weeks, six months, and 12 months postpartum
  A survey designed to provide an overview of individual satisfaction with a program or intervention

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Newport Hospital, Newport, Rhode Island
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - South County Hospital, Wakefield, Rhode Island
  - Kent Hospital, Warwick, Rhode Island
  - Landmark Hospital, Woonsocket, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected from human subjects and will be shared according to NIH guidelines. The investigators are committed to the sharing of final data, being mindful that the rights and privacy of people who participate in research must be protected at all times. The investigators will make a complete study dataset available for sharing. The investigators will have a description of study dataset, including code books, meta-data related to the dataset, and documented programming code used for creating the final study population, for creating variables, and for conducting all outcomes analyses. The investigators will remain HIPAA compliant, and therefore any datasets resulting from participants will be free of any identifiers that would permit linkages to individual research participants and variables that could lead to deductive disclosure of individual subjects.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 5 years after completion of study
Access Criteria: The investigators will make the data and associated documentation available to users under a data-sharing agreement that provides for commitment to: a) using the data only for research purposes and not to identify any individual participant; b) securing the data using appropriate computer technology; and c) destroying or returning the data after analyses are completed. Timelines for distribution of data will vary depending on any required restrictions as mentioned above. Data may be distributed by a number of electronic methods, including web-based databases, datasets, and spreadsheets, or via electronic media such as compact discs.

REFERENCES:
- [Derived] Nunez SD, Spratt LM, Ware CF, Machado S, Rousseau J, Jackson TL, Buckley J, Magee S, Wohler D, Blosser E, Sales S, Simmons D, Ramos VN, Castillo MM, Murray C, Bailey K, Gutman R, Richardson CR, Grobman WA, Hauspurg A, Miller ES, Tuuli MG, Lewkowitz AK. Protocol for a type 1 hybrid effectiveness implementation trial to evaluate whether a technology-based collaborative care model is non-inferior to remote blood pressure monitoring on persistent hypertension and preventive care attendance among postpartum people with hypertension. Contemp Clin Trials. 2025 Dec;159:108114. doi: 10.1016/j.cct.2025.108114. Epub 2025 Oct 23. PMID 41139061